CLINICAL TRIAL: NCT03443739
Title: Medical And Psychological Effects of Nineteen Days of Intermittent Religious Fasting for Followers of the Bahá'í Faith- an Observational Study
Brief Title: Effects of Fasting in the Bahá'í Faith
Acronym: BF
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Universität Münster (Other)
Responsible Party: Principal Investigator, Andreas Michalsen, Clinical professor, Charite University, Berlin, Germany
Other Study IDs: Bahá'í fast
Record Dates: First submitted 2018-02-17; First posted 2018-02-23 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Health Behavior; Healthy
Keywords: Intermittent Fasting; Religious Fast; Bahá'í; Hydration; Calorimetry; Microdialysis; circadian clock; circadian rhythm; spirituality; self-efficacy
MeSH Terms: conditions — Health Behavior; Intermittent Fasting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood, urine
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Intermittent Fasting — Intermittent Fasting with abstinence from food and drink daily from sunrise to sunset for nineteen consecutive days in March 2018

SUMMARY:
The aim of the study is to find out the effects a specific religious fast (i.e. Bahá'í fast) has on certain metabolic parameters, hydration, psyche and circadian clock. In a follow-up questionnaire series in 2019 we want to additionally validate a specific questionnaire for Bahai fasting, which was developed in 2018.

DETAILED DESCRIPTION:
Followers of the Bahá'í Faith worldwide follow a yearly fasting tradition, where they fast intermittently for nineteen days. The intermittent fast is defined as abstinence from any food, drink and smoking from sunrise until sunset. These nineteen days are always in March and so do not coincide with climatic extremes in any country worldwide. This makes this kind of fasting a good model to study the psychological and medical effects of intermittent fasting in humans.

ELIGIBILITY:
Inclusion Criteria:

* member of the Bahá'í religious community, Age between 18-69 years, the study participant must be able to understand the instructions given to him by the study personnel, the performance of the religious fast is planned in 2018 (and for the validation of the questionnaire also in 2019)

Exclusion Criteria:

* An interruption of the religious fast is planned for more than five days, pregnant and nursing women, severe internistic condition, eating disorders (anorexia nervosa, bulimia), terminal or severe disease with marked impairments in mobility and vitality, non-existence of email address and Internet Access (because of online questionnaires), severe psychiatric disorder, simultaneous participation in another Trial

Exclusion Criteria for subsample (energy metabolism measurements and microdialysis)

* Body Mass Index <18,0 und >30,9 kg/m2, claustrophobia, clinically relevant haemostaseological conditions or medication, vegan diet, special diet out of medical reasons, current dieting for weight loss, weight loss of more than 2 kg in the month before the study commenced, postsurgical conditions, acute and chronic infections, known drug or alcohol abuse
* additional exclusion criteria for microdialysis (subsample of energy metabolism measurements): allergy to local anaesthetics

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Members of the Bahá'í community residing in Germany
Sampling Method: Non-Probability Sample
Enrollment: 145 (Actual)
Dates: Start 2018-02-19 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Serum Osmolarity | 12 hours
  Measured in subsample of study participants (venous blood sample) osmol/l
In 2019: Validation of new questionnaire | 1 hour
  New questionnaire, developed in 2018, regarding Bahai fasting

SECONDARY OUTCOMES:
Urine Osmolality | 24 hours
  Measured in subsample of participants, in spontaneous Urine sample and 12h/24h Urine samples osmol/kg
Acid-base balance | 5 Minutes
  Measured in subsample of study participants (venous blood sample) Measured with Radiometer, Base excess (mmol/l)

OTHER OUTCOMES:
Questionnaire: HADS (Hospital Anxiety and Depression Score) | 5 Minutes
  Anxiety and depression
Systolic and diastolic blood pressure | 5 Minutes
  Measured in subsample of study participants Measured by clinician, mmHg
BMI | 10 Minutes
  Measured in subsample of study participants Quantitative, kg/m2
Microdialysis | 3 hours
  Measured in subsample of study participants
Indirect calorimetry | 2 hours
  Measured in subsample of study participants
Individual Interview | 30 Minutes, three times during study
  Measured in subsample of study participants
Activation of clock genes | 3 Minutes
  Measured in subsample of study participants Measured in monocytes

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Michalsen, Prof. Dr., Principal Investigator — Charité University Medicine
Locations (1):
- Charité, Berlin, Germany

REFERENCES:
- [Result] Koppold-Liebscher DA, Klatte C, Demmrich S, Schwarz J, Kandil FI, Steckhan N, Ring R, Kessler CS, Jeitler M, Koller B, Ananthasubramaniam B, Eisenmann C, Mahler A, Boschmann M, Kramer A, Michalsen A. Effects of Daytime Dry Fasting on Hydration, Glucose Metabolism and Circadian Phase: A Prospective Exploratory Cohort Study in Baha'i Volunteers. Front Nutr. 2021 Jul 29;8:662310. doi: 10.3389/fnut.2021.662310. eCollection 2021. PMID 34395487
- [Result] Mahler A, Jahn C, Klug L, Klatte C, Michalsen A, Koppold-Liebscher D, Boschmann M. Metabolic Response to Daytime Dry Fasting in Baha'i Volunteers-Results of a Preliminary Study. Nutrients. 2021 Dec 29;14(1):148. doi: 10.3390/nu14010148. PMID 35011024
- [Derived] Steckhan N, Ring R, Borchert F, Koppold DA. Triangulation of Questionnaires, Qualitative Data and Natural Language Processing: A Differential Approach to Religious Baha'i Fasting in Germany. J Relig Health. 2024 Oct;63(5):3360-3373. doi: 10.1007/s10943-023-01929-x. Epub 2023 Oct 25. PMID 37878201
- See also: Results publication 1 — https://www.frontiersin.org/articles/10.3389/fnut.2021.662310/full